CLINICAL TRIAL: NCT07191756
Title: A Retrospective, Multicenter Cohort Study Comparing the Efficacy and Safety of Amphotericin B Versus Isavuconazole for the Treatment of Mucormycosis: Analysis of Institutional Data and Literature Review
Brief Title: Amphotericin B Versus Isavuconazole for Mucormycosis: A Comparative Efficacy and Safety Study
Acronym: AIM
Status: Active, not recruiting | Type: Observational
Sponsor: Qiu Ye (Other)
Collaborators: Guangzhou Medical University (Other)
Responsible Party: Sponsor-Investigator, Qiu Ye, PhD, Guangxi Medical University
Organization: Guangxi Medical University (Other)
Other Study IDs: 2025-AMB-ISA
Record Dates: First submitted 2025-09-17; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Mucormycosis
Keywords: Amphotericin B; isavuconazole; mucormycosis
MeSH Terms: conditions — Mucormycosis | interventions — Amphotericin B; isavuconazole

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Amphotericin B Cohort: Patients with a confirmed diagnosis of mucormycosis who received primary treatment with any formulation of amphotericin B (e.g., liposomal amphotericin B, amphotericin B deoxycholate) during the study period. Treatment details, including dosage and duration, were collected from retrospective review of electronic medical records from three participating hospitals.
  Interventions: Drug: Amphotericin B
- Isavuconazole Cohort: Patients with a confirmed diagnosis of mucormycosis who received primary treatment with isavuconazole during the study period. Treatment details, including dosage and duration, were collected from retrospective review of electronic medical records from three participating hospitals.
  Interventions: Drug: Isavuconazole

INTERVENTIONS:
Drug: Amphotericin B — This is a retrospective observational study. Patients in this cohort received various formulations of amphotericin B as part of their standard medical care.
  Groups: Amphotericin B Cohort
Drug: Isavuconazole — This is a retrospective observational study. Patients in this cohort received isavuconazole as part of their standard medical care.
  Groups: Isavuconazole Cohort

SUMMARY:
Background:

Mucormycosis is a serious but rare fungal infection that requires rapid and effective treatment. The two main antifungal medicines used are amphotericin B and isavuconazole. However, more real-world data is needed to directly compare how well they work and how safe they are for patients.

What is the purpose of this study? The main goal of this research study is to compare the effectiveness and safety of amphotericin B versus isavuconazole in treating mucormycosis. Investigators will look at which medicine leads to better survival rates and fewer serious side effects.

How will the study be done? This is a retrospective study. This means investigators will look back at information that has already been collected. Investigators will analyze data from the medical records of patients who were treated for mucormycosis at three hospitals. Investigators will also review and combine findings from relevant studies published on PubMed.

What will the researchers measure?

Investigators will measure and compare:

How long patients survived after treatment (survival rates).

Whether the infection was successfully cured or controlled (treatment response).

What kinds of side effects (like kidney problems or liver issues) patients experienced with each medicine.

What are the possible benefits of this study? This study will not directly benefit the participants whose records are reviewed. However, investigators hope that what investigators learn will help doctors make better treatment decisions for future patients with mucormycosis by providing clearer evidence on the best choice of medicine.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of mucormycosis based on histopathology, culture, or typical radiographic findings in accordance with established guidelines.
2. Received primary antifungal treatment for mucormycosis with either amphotericin B (any formulation) or isavuconazole for at least 48 hours.
3. Had at least one follow-up assessment after initiation of antifungal therapy to evaluate treatment response.
4. Medical records from the participating hospitals are sufficiently complete for data extraction regarding treatment and outcomes.

Exclusion Criteria:

* Patients who were not treated with amphotericin B or isavuconazole; and patients who did not have mucormycosis.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study will analyze a retrospective cohort of patients with a confirmed diagnosis of mucormycosis who were treated at one of three participating hospitals. The study population will be divided into two groups based on the primary antifungal therapy they received: (1) those who received amphotericin B-based therapy (any formulation), and (2) those who received isavuconazole. Data from eligible patients' medical records will be extracted to form the final study dataset. Additionally, relevant patient data from studies identified via a systematic PubMed literature review may be included to supplement the analysis.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2025-07-21 (Actual); Study Completion 2025-09-25 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From date of diagnosis until the date of death from any cause, whichever occurred first, assessed up to 12 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: Undecided